CLINICAL TRIAL: NCT00939926
Title: Bioequivalence Study of Risperidone 1 mg Tablets of Torrent Pharmaceuticals Limited., India and Risperdal® (Risperidone) 1 mg Tablets of Janssen Pharmaceutical Products, LP, USA, in Healthy Human Adult Subjects, Under Fed Conditions
Brief Title: Bioequivalence Study of Risperidone 1 mg Tablets of Torrent Pharmaceuticals Limited, India and Risperdal® (Risperidone) 1 mg Tablets of Janssen Pharmaceutical Products, LP, USA, in Healthy Human Adult Subjects, Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Other Study IDs: 1120/07
Record Dates: First submitted 2009-07-10; First posted 2009-07-15 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
Objective:

* To assess the bioequivalence of Risperidone 1.0 mg tablets of Torrent Pharmaceuticals Limited., India and Risperdal® (Risperidone) 1.0 mg tablets of Janssen Pharmaceutical Products, LP, USA, in healthy human adult subjects, under fed conditions.

Study Design:

* A randomized, open label, two treatment, two period, two sequence, single dose, crossover study, under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects of either sex between 18-55 years of age (inclusive) have a body mass index (BMI) between 18 and 27 kg/m2.
2. Subjects who had no evidence of underlying disease during screening and whose physical examination was performed within 21 days prior to commencement of the study.
3. Subjects whose screening laboratory values were within normal limits or considered by the Investigator to be of no clinical significance.
4. Informed consent given in written form according to section 11.3 of the protocol.
5. Female Subjects:

   * of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the Investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine contraceptive device, (IUD) or abstinence.
   * postmenopausal for at least 1 year.
   * surgically sterile (bilateral tubal ligation, bilateral oophorectomy,or hysterectomy).

Exclusion Criteria:

1. History or presence of significant:

   * Cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, musculoskeletal, neurological or psychiatric disease.
   * Alcohol dependence, alcohol abuse or drug abuse within past one year.
   * Moderate to heavy smoking (>10 cigarettes/day) or consumption of tobacco products.
   * History of difficulty in swallowing tablets.
   * Clinically significant illness within 4 weeks before the start of the study.
   * Asthma, urticaria or other allergic type reactions after taking any medication.
   * Positive urine drug screening, HIV, hepatitis B & C tests.
   * Any history of hypersensitivity to Risperidone.
2. Participation in any clinical trial within the preceding 12 weeks of study start.
3. Subjects who had:

   * Systolic blood pressure less than 90 mm of Hg or more than 150 mm of Hg.
   * Diastolic blood pressure less than 60 mm of Hg or more than 94 mm of Hg Minor deviations (2-4 mm Hg) at check-in, if any, were acceptable at the discretion of the physician /Investigator.
   * Pulse rate below 50 /min or above 105 /min.
4. Female subjects demonstrating a positive pregnancy screen or currently breast-feeding or whose menstruation cycle coincides with the study dates.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Labs Pvt. Ltd., Bangalore, Karnataka, India